CLINICAL TRIAL: NCT00251641
Title: An Open-Label, Randomized Efficacy and Safety Study of Infliximab Versus Methotrexate in the Treatment of Moderate to Severe Psoriasis
Brief Title: The Effects of Infliximab Versus Methotrexate in the Treatment of Moderate to Severe Psoriasis (Study P04271AM2)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04271
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Results first posted 2009-07-14 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infliximab (Experimental)
  Interventions: Drug: infliximab
- Methotrexate (Active Comparator)
  Interventions: Drug: methotrexate

INTERVENTIONS:
Drug: infliximab — The infliximab dose will be prepared according to the subject's weight (5 mg/kg). Each intravenous (IV) infusion will be administered over a period of not less than 2 hours. The infusion must be given via a separate line using the administration set with a 1.2 micron filter. Subjects will be infused at Weeks 0, 2, 6, 14, and 22.
  Other Names: SCH 215596; Remicade
  Arms: Infliximab
Drug: methotrexate — Methotrexate will be supplied as 2.5 mg tablets. Subjects are to take 15 mg/week orally for the first 6 weeks of the study. Subjects will be advised to take their MTX as a single dose (weekly) on the same day of the week. If subjects randomized to MTX 15 mg/week experience a <25% reduction in PASI score at Week 6 (Visit 4) as compared with Baseline, their MTX dose will be increased to 20 mg/week. Subjects will be treated for 22 weeks.
  Other Names: Trexall; Rheumatrex
  Arms: Methotrexate

SUMMARY:
This is a Phase 3b, randomized, parallel-group, multicenter, active-controlled, open-label study of the efficacy and safety of infliximab compared with methotrexate (MTX) in the treatment of moderate to severe psoriasis in adults who were diagnosed with moderate to severe plaque-type psoriasis for at least 6 months prior to screening (subjects with concurrent psoriatic arthritis may also be enrolled).

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects (>= 18 to 75 years of age) with a diagnosis of moderate to severe plaque-type psoriasis for at least 6 months prior to study screening (subjects with concurrent psoriatic arthritis may also be enrolled).
* Subjects must be eligible for phototherapy or systemic therapy for their psoriasis and must have a Baseline Psoriasis Area and Severity Index (PASI) score of 12 or greater and have at least 10% of their total body surface area (BSA) involved at Baseline.
* Subjects must agree to avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet light sources during the study.
* Subjects must also meet the tuberculosis (TB) eligibility assessment and screening criteria as follows: Have no history of latent or active TB prior to screening; have no signs or symptoms suggestive of active TB upon medical history and/or physical examination; have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study medication; within 1 month prior to the first administration of study medication, either have negative diagnostic TB test results (defined as 2 negative tuberculin skin tests) OR have a newly identified positive diagnostic TB test result (defined as at least 1 positive tuberculin skin tests) during screening in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study medication.
* Subjects must have had a chest x-ray (posterior-anterior and lateral) within 3 months prior to Screening with no evidence of malignancy, infection, fibrosis, or current or old active TB.
* Specific parameters must also be met with regard to screening laboratory test results and liver enzymes in order to be eligible to participate in the study.

Exclusion Criteria:

* Subjects who have non-plaque forms of psoriasis, current drug-induced psoriasis, are pregnant, nursing, or planning pregnancy;
* Subjects previously treated with MTX or infliximab; subjects who are taking specific drugs within the specified time frame prior to Baseline as follows: any therapeutic agent targeted at reducing tumor necrosis factor (TNF) or any biologic, live virus or bacterial vaccinations within 3 months; any systemic medications or treatments that could affect psoriasis or PASI evaluations, or any systemic immunosuppressants or lithium within 4 weeks; any topical medications or treatments that could affect psoriasis or PASI evaluations within 2 weeks. The only allowed topical treatments for psoriasis are shampoos (containing tar or salicylic acid only) and topical moisturizers. Subjects should not use these topical agents during the morning prior to a study visit. Non-medicated shampoos may be used on the morning of a visit.
* Subjects with poor health, including concomitant congestive heart failure (CHF); history of chronic or recurrent infectious disease, as specified; human immunodeficiency virus, hepatitis B, or hepatitis C; demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis; systemic lupus erythematosus; or who have had serious infections (eg, hepatitis, pneumonia, or pyelonephritis], or who have been hospitalized or received IV antibiotics, or who had an opportunistic infection (eg, cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB), or a transplanted organ within specified time frames; or other conditions as specified in the protocol.
* Subjects who have used any investigational drugs within 4 weeks of Screening, who are participating in other clinical studies, staff or family members of study staff are excluded from participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2005-09-01 (Actual); Primary Completion 2008-06-01 (Actual); Study Completion 2008-06-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Barker J, Hoffmann M, Wozel G, Ortonne JP, Zheng H, van Hoogstraten H, Reich K. Efficacy and safety of infliximab vs. methotrexate in patients with moderate-to-severe plaque psoriasis: results of an open-label, active-controlled, randomized trial (RESTORE1). Br J Dermatol. 2011 Nov;165(5):1109-17. doi: 10.1111/j.1365-2133.2011.10615.x. PMID 21910713

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate: Methotrexate (MTX) will be supplied as 2.5 mg tablets. Subjects are to take 15 mg/week orally for the first 6 weeks of the study. Subjects will be advised to take their MTX as a single dose (weekly) on the same day of the week. If subjects randomized to MTX 15 mg/week experience a <25% reduction in PASI score at Week 6 (Visit 4) as compared with Baseline, their MTX dose will be increased to 20 mg/week. Subjects will be treated for 22 weeks.
Period: Overall Study
Arm/Group | Infliximab | Methotrexate
Started | 653 | 215
Completed | 541 | 127
Not Completed | 112 | 88
Not completed — Adverse Event | 80 | 8
Not completed — Lack of Efficacy | 2 | 1
Not completed — Progression of Disease | 0 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Protocol Violation | 10 | 2
Not completed — Did not Meet protocol Eligibility | 2 | 1
Not completed — Switched Treatment | 9 | 63

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Methotrexate | Total
Number analyzed (Participants) | 653 | 215 | 868
Age, Continuous [Mean (Full Range); unit: years] | 44.1 [18 to 78] | 41.9 [18 to 69] | 43.6 [18 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 67 | 282
  Male | 438 | 148 | 586

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index 75 (PASI75) Response at Week 16.
Description: PASI75 response is defined as the proportion of participants who achieved at least a 75% improvement in PASI score from Baseline.
Time Frame: 16 weeks
Population: All subjects who were randomized were included in the efficacy analysis (intent-to-treat [ITT]).
Measure: Number; unit: Proportion of participants
Arm/Group | Infliximab | Methotrexate
Number analyzed (Participants) | 653 | 215
Proportion of participants | 0.78 | 0.42
Statistical Analysis 1: Comparison: Infliximab vs Methotrexate; The treatment comparison for this endpoint was carried at the 4.9% level of significance; Test type: Superiority or Other; p < 0.001, Chi-squared; Pearson's chi-square test

2. Secondary Outcome: PASI75 Response at Week 26
Description: as for outcome 1
Time Frame: 26 weeks
Population: Intent-to-treat
Measure: Number; unit: Proportion of participants
Arm/Group | Infliximab | Methotrexate
Number analyzed (Participants) | 653 | 215
Proportion of participants | 0.77 | 0.31
Statistical Analysis 1: Comparison: Infliximab vs Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared — Multiplicity adjustment was provided using Hochberg test; Pearson's chi-square test

3. Secondary Outcome: Proportion of Participants Who Achieved a Physician's Global Assessment (PGA) Score of Cleared or Minimal at Week 16
Description: PGA is assessed relative to baseline condition and is defined as: clear (100% clear; some residual pinkness or pigmentation: Wornoff's ring may be present), excellent/minimal (75-99% clearing; marked improvement: nearly normal skin texture; some erythema may be present), good (50-74% clearing; moderate improvement: plaque has cleared to point of small scattered papules with normal intervening epidermis), fair (25-49% clearing; slight improvement: decrease in scaling and softening of plaque), poor (0-24% clearing; little or no change in scaling, erythema, or plaque elevation), or worse (worse).
Time Frame: 16 weeks
Population: ITT
Measure: Number; unit: Proportion of participants
Arm/Group | Infliximab | Methotrexate
Number analyzed (Participants) | 653 | 215
Proportion of participants | 0.76 | 0.38
Statistical Analysis 1: Comparison: Infliximab vs Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared — Multiplicity adjustment was provided using the Hochberg test; Pearson's chi-square test

4. Secondary Outcome: Proportion of Participants Who Achieved a PGA Score of Cleared or Minimal at Week 26
Description: as for outcome 3
Time Frame: 26 weeks
Population: ITT
Measure: Number; unit: Proportion of participants
Arm/Group | Infliximab | Methotrexate
Number analyzed (Participants) | 653 | 215
Proportion of participants | 0.73 | 0.28
Statistical Analysis 1: Comparison: Infliximab vs Methotrexate; Test type: Superiority or Other; p < 0.001, Chi-squared — Multiplicity adjustment was provided using the Hochberg test; Pearson's chi-square test

ADVERSE EVENTS:
Groups:
- Infliximab; Methotrexate: Adverse events reported through Week 26 for participants who did not switch treatment at Week 16 and adverse reported through Week 16 for those participants who switched treatment.
- Participants Who Switched From Infliximab to Methotrexate: Adverse events reported for participants who switched from infliximab to methotrexate at Week 16 (including only adverse events with begin dates on or after a switch in treatment).
- Participants Who Switched From Methotrexate to Infliximab: Adverse events reported for participants who switched from methotrexate to infliximab at Week 16 (including only adverse events with begin dates on or after a switch in treatment).
Arm/Group | Infliximab | Methotrexate | Participants Who Switched From Infliximab to Methotrexate | Participants Who Switched From Methotrexate to Infliximab
Serious Adverse Events (participants affected / at risk) | 44/649 | 6/211 | 0/9 | 3/63
Other Adverse Events (participants affected / at risk) | 275/649 | 95/211 | 1/9 | 11/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=649) | Methotrexate (N=211) | Participants Who Switched From Infliximab to Methotrexate (N=9) | Participants Who Switched From Methotrexate to Infliximab (N=63)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
IRIDOCYCLITIS (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MACULAR HOLE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
TYPE IV HYPERSENSITIVITY REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEBRILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYME DISEASE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FOCAL NODULAR HYPERPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TESTICULAR NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVARIAN HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=649) | Methotrexate (N=211) | Participants Who Switched From Infliximab to Methotrexate (N=9) | Participants Who Switched From Methotrexate to Infliximab (N=63)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 (9) | 11 (27) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 21 (22) | 17 (34) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 21 (30) | 20 (77) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 26 (28) | 19 (39) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 70 (139) | 0 (0) | 0 (0) | 5 (10)
NASOPHARYNGITIS (Infections and infestations) | 119 (157) | 40 (46) | 0 (0) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 41 (54) | 12 (15) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 66 (111) | 31 (74) | 0 (0) | 5 (7)
EPIDIDYMITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 39 (50) | 4 (4) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must provide sponsor w/ review copies of abstracts or manuscripts for publication that report any results of the study, 45 days before submission for publication or presentation. The sponsor shall have the right to review/comment on the material. If the parties disagree about the appropriateness of the material, PI must meet with sponsor's representatives before submission for publication, for the purpose of making good faith efforts to discuss and resolve any issues of disagreement.